CLINICAL TRIAL: NCT02041793
Title: A Prospective Randomized Controlled Trial Comparing Laparoscopic Versus Endoscopic Drainage for Pseudocyst of the Pancreas
Brief Title: Laparoscopic Cystogastrostomy Versus Endoscopic Cystogastrostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr Virinder Kumar Bansal, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICMR-PP 5/10
Record Dates: First submitted 2013-07-10; First posted 2014-01-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Pancreatic Pseudocyst
Keywords: Acute pancreatitis; Pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst; Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic cystogastrostomy (Active Comparator): Laparoscopic cystogastrostomy will be performed by using a stapled cystogastrostomy
  Interventions: Procedure: Laparoscopic cystogastrostomy
- Endoscopic cystogastrostomy (Active Comparator): Endoscopic cystogastrostomy or cystoduodenostomy will be performed either under direct endoscopic or endosonography guidance.
  Interventions: Procedure: Endoscopic cystogastrostomy

INTERVENTIONS:
Procedure: Laparoscopic cystogastrostomy — Patients undergo drainage of pseudocyst by laparoscopic technique
  Arms: Laparoscopic cystogastrostomy
Procedure: Endoscopic cystogastrostomy — Endoscopic cystogastrostomy or cystoduodenostomy will be performed either under direct endoscopic or endosonography guidance
  Arms: Endoscopic cystogastrostomy

SUMMARY:
This study is a randomized controlled trial comparing Laparoscopic and endoscopic drainage for pseudocyst of the pancreas secondary to acute pancreatitis. The primary outcome measure will be resolution of the pseudocyst by the intended treatment within 4 weeks. The secondary outcomes will be complications, recurrence and cost analysis between the two methods.

DETAILED DESCRIPTION:
This study will be conducted in the Department of Surgical Disciplines and Department of Gastroenterology, All India Institute of Medical Sciences, New Delhi. Patients with pancreatic pseudocyst will be randomized to two groups-

Group I- Laparoscopic management of the pseudocyst Group II- Endoscopic management of the pseudocyst

Patients will be randomized using computer generated randomized numbers in sealed envelopes to ensure concealed allocation with block randomization. The details of patients who do not meet inclusion criteria and those who refuse consent and reason for refusal of consent will also be noted. Refusal for consent for inclusion in the study will not hamper the treatment of these patients in anyway. The patients will be evaluated prospectively. CONSORT guidelines will be followed.

Preoperative Data

The details regarding demographic profile of the patient i.e. age/ sex/ body mass index (BMI) and clinical features will be noted. The duration and presenting complaint for pseudocyst and history regarding the acuteness of underlying pancreatic disease will be noted. The etiology of pancreatitis will be noted. Patients will be examined thoroughly and the characteristic features of the pseudocysts, the size and the site (head, body or tail of the pancreas) will be noted. The American Society of Anesthesiologists (ASA) grading of the patient will also be done.

Pre-operative Investigations

Preoperative investigations will include hemogram, liver function tests, serum electrolytes, serum amylase, serum lipase, kidney function tests, chest X-ray and electrocardiogram. Ultrasound of the abdomen, and contrast enhanced computer tomography (CECT) will be done for proper localization, size, wall characteristics, presence or absence of pseudoaneurysm and relationship of the cyst with the surrounding structures. Magnetic Resonance Imaging (MRI) will be done to asses the relative amount of necrotic debris within the cyst, if required. An Endoscopic ultrasound will be done at the discretion of the gastroenterologist for planning endoscopic drainage of the pseudocyst.

A clinical case record (CRF) form will be filled with all the relevant details.

INTERVENTION TECHNIQUE

Laparoscopic Cystogastrostomy

Pre-operative Preparation

One dose of injection cefoperazone 1000 mg + sulbactam 1000 mg after skin test, one dose of metronidazole 500 mg and Amikacin 1000 mg will be given intravenously as prophylaxis pre-operatively at the time of induction of anesthesia. The antibiotics will be continued for 3 days after surgery. A 14 Fr Foley's catheter will be placed pre-operatively after induction of anesthesia.

Operative Procedure

Patient will be placed in Lloyd-Davis position with both upper limbs by side of the patient. General anesthesia with or without supplementation with spinal anesthesia will be given to all patients. A 12 mm camera port at umbilicus, one 5 mm port in the left pararectal region, one 12 mm port in the right pararectal area at the level of umbilicus and the fourth port in the epigastric region for puncturing and aspirating the pseudocyst. 2-3 ml of 0.25% bupivacaine will be infiltrated at each port site for local anesthesia before port placement. Pneumoperitoneum will be created using veress needle. The first port will be inserted in a closed manner and directed towards the upper abdomen. The bulge of the pseudocyst on the posterior wall of the stomach will be identified and access to the posterior gastric wall will be established through an anterior gastrotomy (2 -2.5 cm) created with the help of harmonic shears/monopolar hook knife. A long needle will be introduced to confirm the location of the pseudocyst and to sample the fluid. A bariatric port will be introduced through the posterior wall of the stomach into the cyst and its contents aspirated. The cyst will then be irrigated through the port and debris cleared. The cystogastrostomy stoma will be made with endostapler (Ethicon Endo-surgery, Cincinnati). Gastrotomy will be closed in two layers with intracorporeal suturing. Cholecystectomy will be done if necessary using the standard four port technique. A 16 F drain will be placed in the subhepatic space.

Details of any associated procedures like cholecystectomy, laparoscopic CBD exploration or any other procedure will be recorded and details noted thereof.

Endoscopic Cystogastrostomy

Preprocedural preparation

One dose of injection cefoperazone 1000 mg + sulbactam 1000 mg after skin test will be given intravenously as prophylaxis before the procedure and will be continued for up to 3 days after the procedure or as required.

Procedure

The ideal site of puncture will be determined by the site of maximum bulge on the posterior gastric wall. A needle knife will be used to puncture into the gastric or cyst wall with the help of electrocoagulation. A gush of cyst fluid will be encountered when the cyst is entered. A guide wire will be then passed through the needle knife. A balloon will be used to dilate the opening up to 15 mm without cutting. One 10 Fr plastic double pigtail stent will be placed into the pseudocyst. The stent will be removed three months later. If there is no bulge on endoscopic view, cystogastrostomy will be done under endoscopic ultrasonography guidance.

In the presence of necrotic debris if a patient develops fever, a repeat procedure will be done within three days. An 8.8 mm diameter, size forward viewing endoscope will be used to enter the cavity. The cavity will be lavaged with saline and loose necrotic tissue will be removed with snare or basket.

Operative data will be recorded in a preformed proforma on port placements, mode of gastrotomy, location of the pseudocyst, operation time, associated procedures performed, conversion to open, any intraoperative complication and other intra-operative details. Reasons for conversion to open and procedure performed after conversion will also be recorded. Data regarding endoscopic procedure will also be recorded in a prestructured proforma on the technique, mode of gastrotomy, procedure time, any complication encountered during the procedure and other intraprocedural details. The number of procedures and hospital stay will be recorded.

Details of any associated procedures like endoscopic retrograde cholangiopancreaticography (ERCP) or Common bile duct (CBD) stone removal will be recorded. An ERCP will not be done routinely prior to drainage to find out any communication of the cyst with main pancreatic duct (MPD). In patients with recurrence within four weeks an ERCP will be done to rule out ductal communication and a pancreatic stent will be placed if a fistula is found in both surgical and endoscopic groups.

Post intervention Evaluation

Data regarding post operative/post endoscopic recovery and complications such as bleeding, wound infection, haematemesis, fever, intra abdominal collection and any drainage performed will be collected. Post operative/post procedural amylase levels and ultrasound findings will also be recorded.

Hospital Stay

Post procedure hospital stay would be recorded in days. Follow up

All patients will be followed up in the post operative period for at least 3 months. The first follow up will be at seven days, then at 4 weeks and then 3 months after surgery. An ultrasound will be done at each follow up to look for cyst recurrence or any other intra-abdominal problem. A note of any additional procedures or admissions after the index intervention will be made.

Cost of procedure

This includes both direct and indirect costs incurred by the patient and the hospital for the procedure.

Statistical analysis

The data will be entered into Microsoft excel software and will be analyzed by using Statistical Package for the Social Sciences (SPSS) software version 15. The statistical method applied will be student t-test/ Mann Whitney U test, whichever is applicable to compare the continuous data between the two groups and the categorical variables will be compared using Chi - Square test/ Fisher exact test. A P-value of <0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

Symptomatic patients with pseudocyst of size more than 6 cm, more than 6-8 weeks duration after an attack of acute pancreatitis.

Exclusion Criteria:

* Patients with chronic pancreatitis associated pseudocyst.
* Patients who have undergone any form of intervention previously
* Patients with significant co-morbidities
* Patients unfit for general anesthesia
* Bleeding disorders
* Patients refusing consent
* Patients having significant necrotic debris not considered fit for endoscopic drainage. The presence of necrotic debris will be assessed by ultrasound of the abdomen and if required magnetic resonance imaging. The volume of the cyst and that of necrotic debris will be calculated and significant debris will be defined as >30% of debris volume/volume
* Presence of a pseudoaneurysm

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Resolution of Pseudocyst | 4 weeks
  resolution on imaging

SECONDARY OUTCOMES:
Adverse Events | 4 weeks
  Bleeding, sepsis, chest complications and other important events in the post procedure period requiring prolonged stay and /or repeat procedure
Cost per patient | 4 weeks
  Cost effectiveness to be calculated from the average cost per patient and the number of successful outcomes.
Recurrence rate of pseudocyst | 3 months
  development of new pseudocyst

CONTACTS AND LOCATIONS:
Overall Officials: Virinder K Bansal, MS, Principal Investigator — All India Institute of Medical Sciences; Pramod K Garg, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Aljarabah M, Ammori BJ. Laparoscopic and endoscopic approaches for drainage of pancreatic pseudocysts: a systematic review of published series. Surg Endosc. 2007 Nov;21(11):1936-44. doi: 10.1007/s00464-007-9515-2. Epub 2007 Aug 24. PMID 17717626